CLINICAL TRIAL: NCT00339885
Title: Mapping Genes for Type 2 (Non-Insulin Dependent) Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995030; OH95-HG-N030
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Genetic Variation; Diabetes
Keywords: Monogenic Diabetes; Type 2 Diabetes Mellitus; QTL
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood DNA, Adipose, Muscle, Fibroblast, Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (16):
- AADM: Family and Population based individuals
- Action-LADA: Population based individuals
- D2D 2004: Population based individuals
- DIAGEN (Dresden Biobank): Population based individuals
- FINRISK 1987: Population based individuals
- FINRISK 2002: Population based individuals; Test DNA
- Fusion 1: Affected-sib pair (ASP) families and elderly controls
- Fusion 2: 275 Replication ASP Families; Trios
- Fusion 3: Siblings of FUSION1 families; Spouses, Offspring of 291 FUSION 1 families; Spouses, Offspring of Elderly Controls; Other F1 relatives
- Fusion 4/5: Spouses, Offspring of FUSION 1 and 2 Families
- FUSION Finnish Groups: Family and Population based (including METSIM and DR's EXTRA): Tissue samples
- Health-2000: Population based individuals
- HUNT 2: Population based individuals
- METSIM: Population based individuals
- Savitaipale: Population based individuals
- UEF - Laakso: Monogenic disease individuals and family members

SUMMARY:
The aim of the project is to positionally clone susceptibility genes for NIDDM. Patients will be ascertained in Finland from previous health surveys and hospital discharge records. Approximately 400 affected sib pairs will be collected. Families will be chosen who have, at most, one parent with NIDDM no history of IDDM. A clinical examination will be undertaken on family members and blood drawn for DNA isolation. Covariates such as body weight, blood pressure, lipid levels and urinary albumin will also be measured. The unaffected spouse and children of a subset of probands will be invited to undergo a frequently-sampled intravenous glucose tolerance test (FSIGT) to measure parameters of pancreatic function and peripheral insulin resistance (IR). A number of unrelated elderly non-diabetic subjects will also be identified to conduct a population-based association analysis.

The FSIGT analysis will be performed in Los Angeles. The DNA will be shipped to Bethesda where a total genomic scan will be performed using semi-automated fluorescence-based genotyping technology. Data from Bethesda, Los Angeles and Finland will be sent to Ann Arbor where parametric and non-parametric methods will be used to analyse both discrete traits such as NIDDM and intermediate traits like IR....

DETAILED DESCRIPTION:
The Finland-United States investigation of NIDDM (FUSION) study is a long-term effort to

identify susceptibility genes for Type 2 diabetes (T2D) and associated quantitative traits. This

involves the phenotyping and DNA analysis of thousands of individuals living in Finland, utilizing a study design that was originally based on affected sib pairs. The majority of these samples have already been subjected to a genome scan using microsatellite markers and the original FUSION samples. Additionally, thousands of other northern European cases and controls have been subjected to genome-wide association (GWA) analysis and/or fine mapping as part of the FUSION study. More recently, the opportunity provided by the lowered sequencing costs have allowed targeted and/or whole genome sequencing of many of these individuals.

ELIGIBILITY:
* No eligibility criteria listed.

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A large majority of the sample population resides in various parts of Finland and are of Finnish descent. The Finnish population provides an ideal basis for studies of complex genetic diseases such as T2D due to its relative genetic and environmental homogeneity, excellent data sources, and a population strongly supportive of biomedical research. Individuals with or without diabetes (type2 or monogenic forms of diabetes) have been collected.
Sampling Method: Non-Probability Sample
Enrollment: 32379 (Actual)
Dates: Start 1996-06-01 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
T2D status, quantitative traits measurements | ongoing
  Association testing

CONTACTS AND LOCATIONS:
Overall Officials: Lori Bonnycastle, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (4):
- Finland (2):
  - Natl Inst for Health & Welfare (THL), Helsinki
  - Research Ethics Committee of Hospital District of Northern Savo, Kuopio
- Norway (2):
  - University of Tromso, Tromsø
  - Norwegian U of Science & Technology, Trondheim